CLINICAL TRIAL: NCT04448951
Title: Immune Homeostasis in Patients With Sepsis and Septic Shock: a Single Center Observational Study
Brief Title: Immune Homeostasis in Sepsis and Septic Shock
Acronym: IMHOTEP
Status: Recruiting | Type: Observational
Sponsor: Charles University, Czech Republic (Other)
Responsible Party: Principal Investigator, Thomas Karvunidis, Principal investigator, Charles University, Czech Republic
Other Study IDs: IMHOTEP
Record Dates: First submitted 2020-06-23; First posted 2020-06-26 (Actual); Last update posted 2024-08-21 (Actual); Status verified 2024-08

CONDITIONS: Sepsis; Immunologic Paralysis; Immunologic Suppression; Immune Deficiency
Keywords: sepsis; septic shock; immune response; immunoparalysis; transcriptomics; flow-cytometry; immunomodulation
MeSH Terms: conditions — Sepsis; Immunologic Deficiency Syndromes; Shock, Septic | interventions — Gene Expression Profiling; Flow Cytometry; Cytokines

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples With DNA — peripheral blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- sepsis/septic shock: target population
  Interventions: Other: transcriptomics; Other: flow-cytometry; Other: cytokines
- non-septic critically ill: demographically-matched control group
  Interventions: Other: transcriptomics; Other: flow-cytometry; Other: cytokines
- healthy control: control group
  Interventions: Other: transcriptomics; Other: flow-cytometry; Other: cytokines

INTERVENTIONS:
Other: transcriptomics — transcriptomics
Other: flow-cytometry — peripheral blood myeloid cells and lymphocytes flow-cytometry
Other: cytokines — peripheral blood cytokine analysis

SUMMARY:
Detailed description of immune response and its dynamics in sepsis and septic shock patiens by means of transcriptomics, flow-cytometry and cytokine analysis.

ELIGIBILITY:
Inclusion Criteria:

* sepsis/septic shock (SEPSIS-3)
* age ≥18
* informed consent
* inclusion within first 24hrs after development/diagnosis of septic shock

Exclusion Criteria:

* disagreement of the patient or legal representative with the entry into the study
* patients with primary or secondary immunodeficiency
* presence of active haematological malignancy or an active non-haematological malignancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: sepsis/septic shock according SEPSIS-3 definition
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2025-08-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Immune response description - flow cytometry | 2024 - 2026
  Detailed description of immune response analyzed by mean of flow cytometry
Immune response description - transcriptomics | 2024 - 2026
  Detailed description of immune response analyzed by mean of transcriptomic analysis
Immune response description - ELISA | 2024 - 2026
  Detailed description of immune response analyzed by mean of ELISA

SECONDARY OUTCOMES:
Diagnostic "immune status" panel | 2026 - 2028
  Diagnostic tool for immune status assessment

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Karvunidis, MD, PhD, Principal Investigator — Carles University Teaching Hospital and Faculty of Medicine in Pilsen, Pilsen, Czech Republic
Locations (1):
- Medical ICU, 1st Dept. of Internal Medicine, Teaching Hospital in Pilsen, Pilsen, Česká Republika, Czechia